CLINICAL TRIAL: NCT00522015
Title: Rivastigmine (Exelon®) for Treatment of Dementia in Patient With Progressive Supranuclear Paresis Open Label Phase 2 Study
Brief Title: Efficacy Study for Treatment of Dementia in Progressive Supranuclear Palsy
Acronym: psp
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Professor Dr. Berg, University hospital of Tuebingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIVA; eudraCT no: 2006-006166-42
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Last update posted 2008-02-18 (Estimated); Status verified 2007-08

CONDITIONS: Progressive Supranuclear Palsy; Dementia
Keywords: PSP; dementia; neuropsychology; treatment
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Dementia | interventions — Rivastigmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator): patients take 6 mg rivastigmine daily, if well tolerable increase to 12 mg rivastigmine maximum daily
  Interventions: Drug: rivastigmine

INTERVENTIONS:
Drug: rivastigmine — rivastigmine 6 mg up to 12 mg daily; Taken in two doses from 3 mg to 6 mg Rivastigmine twice a day
  Other Names: Exelon

SUMMARY:
to show that

1. patients improve and stabilize after 12 -24 week treatment with rivastigmine in memory function
2. use of rivastigmine has a positive effect on apathy in PSP patients
3. therapy with rivastigmine has a no positive benefit on speech and overall results of the MMST
4. changes in motor activity are associated with changes in language and overall results of the in MMST

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PSP
* willingness to participate in the study
* informed consent
* ability to speak
* no further CNS diseases
* written informed consent
* stable state of health
* ability to give informed consent, will checked by an independent physician

Exclusion Criteria:

* alcohol abuses
* acute psychosis
* pregnancy or lactation
* known previous drug reaction or hypersensitivity of rivastigmine or other carbamate derivatives
* liver failure
* known sick sinus syndrome or excitation disturbance
* known ulcus ventriculi or duodenal ulcer
* known asthma or COPD
* seizures
* renal failure

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-12; Study Completion 2010-02

PRIMARY OUTCOMES:
improvement in neuropsychological assessments for memory and executive function, e.g. tested by "Tower of London Test, CERAD Battery and Logical Memory Test (WMSR)" | 6 month

SECONDARY OUTCOMES:
changes in speech function and improvement of quality of life | 6 Month

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Berg, Doctor, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University of Tuebingen, Tübingen, Baden-Wurttemberg, Germany